CLINICAL TRIAL: NCT01030107
Title: Sleep Duration and Pediatric Overweight: the Role of Eating Behaviors
Brief Title: Effects of Sleep Duration on Eating and Activity Behaviors
Status: Completed | Type: Observational
Sponsor: The Miriam Hospital (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Other Study IDs: 1-08-JF-17
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2011-04

CONDITIONS: Sleep; Obesity
Keywords: sleep; obesity; children; eating behaviors; activity; leptin; ghrelin
MeSH Terms: conditions — Obesity; Feeding Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 ml of whole blood drawn at each of 3 assessments
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with Insufficient Sleep: Children who sleep approximately 9-10 hours/night
  Interventions: Behavioral: Increase Sleep; Behavioral: Decrease Sleep

INTERVENTIONS:
Behavioral: Increase Sleep — Children are asked to increase their sleep by approximately 1 1/2 hours/night for 1 week.
Behavioral: Decrease Sleep — Children are asked to decrease their sleep by approximately 1 1/2 hours/night.

SUMMARY:
The purpose of the proposed study is to determine whether the amount children sleep is associated with changes in hormones, hunger, motivation to eat, and food intake. Fifty children 8-11 years old who sleep 9-10 hours per night will be enrolled for a 3-week study. For 1 week each, children will be asked to sleep their typical amount, increase their sleep by 1-½ hours, and decrease their sleep by 1-½ hours. Half of the children will be asked to increase their sleep first and half to decrease their sleep first. During each week, the following will be gathered: sleep duration (measured by actigraphy, which is a small device that measures sleep), levels of hormones measured through blood draws, self-reported hunger and appetite, food intake (measured by 3 days of 24-hour recall), how motivated children are to eat (measured using a computer activity), and child height and weight. We believe that when children sleep less they will show changes in hormones associated with hunger and appetite, report being hungrier, be more motivated to eat, and eat more food.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-11 years old
* BMI for age and gender > 5th percentile (but no greater than 100% overweight)
* Sleep approximately 9-10 hours nightly
* Attend elementary school
* Like at least 1 food and 1 activity used in the reinforcement paradigm
* Able to understand and complete the reinforcement paradigm

Exclusion Criteria:

* Existence of a diagnosable sleep disorder
* Medical or psychiatric condition that could influence sleep or weight
* Onset of menarche
* Inability to complete study materials, including diagnosed disabilities
* Dietary restrictions/allergies to foods used in the study that preclude them from study participation

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children ages 8-11 years old recruited from Southeastern New England.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
absolute reinforcing value of food as compared to sedentary activities | after 1 week of typical sleep duration, after 1 week of decreased sleep duration, after 1 week of increased sleep duration

SECONDARY OUTCOMES:
plasma levels of leptin and ghrelin | after 1 week of typical sleep duration, after 1 week of decreased sleep duration, after 1 week of increased sleep duration
caloric intake | after 1 week of typical sleep duration, after 1 week of decreased sleep duration, after 1 week of increased sleep duration
levels of physical activity | after 1 week of typical sleep duration, after 1 week of decreased sleep duration, after 1 week of increased sleep duration
subjective ratings of hunger and appetite | after 1 week of typical sleep duration, after 1 week of decreased sleep duration, after 1 week of increased sleep duration

CONTACTS AND LOCATIONS:
Overall Officials: Chantelle N Hart, PhD, Principal Investigator — The Miriam Hospital/Alpert Medical School of Brown University
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Hart CN, Spaeth AM, Egleston BL, Carskadon MA, Raynor HA, Jelalian E, Owens JA, Considine RV, Wing RR. Effect of changes in children's bedtime and sleep period on targeted eating behaviors and timing of caloric intake. Eat Behav. 2022 Apr;45:101629. doi: 10.1016/j.eatbeh.2022.101629. Epub 2022 Mar 26. PMID 35390756
- [Derived] Hart CN, Carskadon MA, Considine RV, Fava JL, Lawton J, Raynor HA, Jelalian E, Owens J, Wing R. Changes in children's sleep duration on food intake, weight, and leptin. Pediatrics. 2013 Dec;132(6):e1473-80. doi: 10.1542/peds.2013-1274. Epub 2013 Nov 4. PMID 24190680
- See also: Weight Control and Diabetes Research Center — http://www.weightresearch.org